CLINICAL TRIAL: NCT03555929
Title: Impact on Sensitivity and Motor Block Duration of an Intravenous Dexamethasone Injected 90 Min After Making an Axillary Block With Mepivacaine. A Prospective, Randomized, Placebo-controlled Study
Brief Title: Impact on Sensitivity and Motor Block Duration of an Intravenous Dexamethasone an Axillary Block With Mepivacaine.
Acronym: DEXA-rescue
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P170701J; 2017-004164-35 (EudraCT Number)
Record Dates: First submitted 2018-03-16; First posted 2018-06-14 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2018-03

CONDITIONS: Hand Wound; Wrist Wound; Forearm Wound; Hand Fracture; Wrist Fracture; Forearm Fracture
Keywords: Axillary block; Dexamethasone; anesthesia
MeSH Terms: conditions — Hand Injuries; Wrist Injuries; Wrist Fractures | interventions — Dexamethasone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Experimental): Dexamethasone 8 mg/2cc I.V. 90 minutes after axillary block
  Interventions: Drug: Dexamethasone
- Normal saline (Placebo Comparator): Normal saline 2cc I.V., 90 minutes after axillary block
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexamethasone — 80 minutes after achievement of axillary block, if the surgery is not ended, patients will be randomly assigned to one of the two groups : DEXA or Control. Injection will be done 90minutes after achievement of axillary block.
  Arms: Dexamethasone
Drug: Normal saline — 80 minutes after achievement of axillary block, if the surgery is not ended, patients will be randomly assigned to one of the two groups : DEXA or Control. Injection will be done 90minutes after achievement of axillary block.
  Arms: Normal saline

SUMMARY:
Intravenous dexamethasone is used to increase the duration of analgesia of interscalene bloc for shoulder surgery: it extends from 11h to 23h the sensitivity block in shoulder area. However, the time of dexamethasone intravenous injection has not been studied. In all studies, dexamethasone was injected right after the achievement of loco regional anesthesia.

The main objective is to demonstrate that intravenous injection of dexamethasone delayed at 90 minutes in patients who received an axillary block with mepivacaine prolongs the duration of the motor block by 40 minutes.

DETAILED DESCRIPTION:
In orthopedic surgery, most of procedures are made under loco regional anesthesia. For a surgery of hand, wrist or forearm, an axillary block is made to obtain an insensitivity (sensitivity block) and an unability to move from elbow to fingers (motor block). Depending on the duration of surgery, less or more than 2 hours, a choice of anesthetic has to be made. For short surgeries, mepivacaine is taken on, but for longer ones, local anesthetics like ropivacaine or levo bupivacaine are recommended. Nevertheless, once surgery started, there isn't any possibility to extend the anesthesia duration in case of an unexpected increase of surgery length. A general anesthesia will therefore be required.

Intravenous dexamethasone is used to increase the duration of analgesia of interscalene bloc for shoulder surgery: it extends from 11h to 23h the sensitivity block in shoulder area(1). However, the time of dexamethasone intravenous injection has not been studied. In all studies, dexamethasone was injected right after the achievement of loco regional anesthesia.

The investigator hypothesized that intravenous dexamethasone could extend anesthetic duration of a mepivacaine axillary block (motor and sensitivity block length) even though dexamethasone was injected 90 min after the achievement of block and could be a good option in case of an unexpected extended surgery.

In orthopedic surgery, most of procedures are made under loco regional anesthesia. For a surgery of hand, wrist or forearm, an axillary block is made to obtain an insensitivity (sensitivity block) and an unability to move from elbow to fingers (motor block). Depending on the duration of surgery, less or more than 2 hours, a choice of anesthetic has to be made. For short surgeries, mepivacaine is taken on, but for longer ones, local anesthetics like ropivacaine or levo bupivacaine are recommended. Nevertheless, once surgery started, there isn't any possibility to extend the anesthesia duration in case of an unexpected increase of surgery length. A general anesthesia will therefore be required.

Intravenous dexamethasone is used to increase the duration of analgesia of interscalene bloc for shoulder surgery: it extends from 11h to 23h the sensitivity block in shoulder area(1). However, the time of dexamethasone intravenous injection has not been studied. In all studies, dexamethasone was injected right after the achievement of loco regional anesthesia.

The investigator hypothesized that intravenous dexamethasone could extend anesthetic duration of a mepivacaine axillary block (motor and sensitivity block length) even though dexamethasone was injected 90 min after the achievement of block and could be a good option in case of an unexpected extended surgery.

52 patients will be randomly assigned to two groups:

* DEXA: dexamethasone 8 mg/2cc I.V. 90 minutes after axillary block
* Control: Normal saline 2cc I.V., 90 minutes after axillary block These patients will be recruited during the anesthesia interview from 1 hospital, with 5 surgeons performing the surgeries and 15 anesthetists performing the axillary block

  1. After written consent, all patients will have their surgery under regional anesthesia only provided by the axillary block, with mepivacaine 1.5% 25cc.
  2. Time of complete motor and sensitivity block will be monitored and recorded
  3. 80 minutes after achievement of axillary block, if the surgery is not ended, patients will be randomly assigned to one of the two groups : DEXA or Control
  4. Injection will be done 90minutes after achievement of axillary block
  5. Monitoring of motor block and sensitivity block recovery will be done :

     * during the surgery by nurse and surgeon
     * after the surgery in recovering room by nurses each 15min.
  6. Patients will be called on post operative day one for pain evaluation and detection of adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Women or men should be operated on hand, wrist or forearm for an elective surgery or emergency surgery
* The surgery will be provided under axillary block, a loco regional anesthesia made under ultrasonography with mepivacaine.
* Women of childbearing/reproductive potential must have effective contraceptive method defined by a hormonal method or an intrauterine device (IUD) or surgical sterilization of the patient or her partner,
* Patients must have French state medical insurance (Patients adhering to Social Security),
* Patients providing the investigator with a signed informed consent

Exclusion Criteria:

* Age under 18yrs
* Pregnant or breastfeeding
* Brachial plexus neuropathy
* Hand or forearm injury with nerve injury (unsensitivity or paralysis)
* Other local anesthetic used: lidocaine, ropivacaine, levo bupivacaine
* Planned general anesthesia in association with loco regional anesthesia
* Diabetes
* Current infection on surgical area, puncture area or general bacterial or viral infection.
* Vaccination with attenuated vaccine in the current month
* Porphyry
* Severe hemostasis trouble
* Any contraindication to mepivacaine/axillary block anesthesia, severe heart rate trouble requesting pacemaker (BAVII, BAV3) and uncontrolled epilepsy
* Routine use of systemic corticosteroid or opioid medication
* Known local anesthetics/mepivacaine allergy
* expected duration of surgery less than 60 minutes
* evolving virosis (hepatitis, herpes, shingles and chickenpox)
* Psychotic states not controlled by treatment
* Dexamethasone (Mylan 4 mg/1 mL) allergy or intolerance
* Patient refusal
* Incapacity to consent: Any disease that may invalidate the understanding of protocol information and informed consent.
* Participation to an other study
* Patient under trusteeship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-16 (Actual)

PRIMARY OUTCOMES:
Duration of motor block | within 3 hours after intervention.
  The evaluation of the appearance of the motor block is done by a neurological examination of the anesthetized hand and forearm every 5 minutes after injection of the local anesthetic during 20 minutes During the intervention, the reappearance of a movement of the hand or forearm is signaled by the surgeon at the request of the anesthetist and corresponds to the end of the motor block.
  After the intervention, a neurological examination is performed every 15 minutes in a recovery room until the appearance of the first movement of the hand

SECONDARY OUTCOMES:
Duration of sensitivity block defined as the time between the performance of sensitivity block and appearance of paresthesic or the first analgesia request. | within 3 hours (for outcome measure 1) (end of intervention for 2 and 3) and at 24 hours after the intervention
Sedation or general anesthesia request | within 3 hours (for outcome measure 1) (end of intervention for 2 and 3) and at 24 hours after the intervention
Pain scores in recovering room | within 3 hours (for outcome measure 1) (end of intervention for 2 and 3) and at 24 hours after the intervention
Adverse effects in next 24 hours | within 3 hours (for outcome measure 1) (end of intervention for 2 and 3) and at 24 hours after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Avicenne, Bobigny, France